CLINICAL TRIAL: NCT04180189
Title: SLEEP - An Intervention With Weighted Blankets for Children With Attention Deficit Hyperactivity Disorder (ADHD) and Sleep Problems
Brief Title: An Intervention With Weighted Blankets for Children With ADHD and Sleep Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halmstad University (Other)
Responsible Party: Principal Investigator, Ingrid Larsson, RN, PhD, Associated Professor, RN, PhD, Associate professor, Halmstad University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1SLEEP
Record Dates: First submitted 2019-11-21; First posted 2019-11-27 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Adhd; Sleep Disturbance
Keywords: children; non-pharmacological intervention; ADHD; sleep
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weighted fiber blanket (Active Comparator): Using a weighted blanket
  Interventions: Other: Weighted fiber blanket
- Regular fiber blanket (Placebo Comparator): Using a specially designed fiber blanket without extra weight.
  Interventions: Other: Weighted fiber blanket

INTERVENTIONS:
Other: Weighted fiber blanket — Using weighted blanket for four weeks

SUMMARY:
The aim of the study is to evaluate a sleep intervention with weighted blankets for children with ADHD and sleep problem regarding health-related outcomes, sleep, and cost-effectiveness.

The study is an RCT with cross-over design. The participants will be randomized to start with an active or placebo blanket, and then change blankets during the 16 week study period.

DETAILED DESCRIPTION:
There is limited evidence about health outcomes or health-economic benefits of sleep interventions with weighted blankets for children with neuropsychiatric syndromes (NPS).

The aim of the study is to evaluate a sleep intervention with weighted blankets for children with ADHD and sleep problem regarding health-related outcomes, sleep, and cost-effectiveness.

The participants, n=100 children between 6 and 13 years old, will be recruited from the ADHD unit in Child and Adolescent Mental Health Service (CAMHS) and randomly assigned into two groups: Fiber Weighted Blankets (intervention 1) and Control Blankets (controls).

The children will use each blanket respectively for 4 weeks, then change blankets. A long term follow-up will be conducted 16 weeks from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with ADHD with sleep problems (defined by screening instrument). -
* Being a patient at child and adolescent mental health service (CAMHS) in Region Halland, Sweden.
* Parents and children should understand (written and spoken) Swedish language.

Exclusion Criteria:

* Already used weighted blankets as a sleep intervention,
* If they have received a new prescription or change of pharmacological treatment for sleep problems

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency | 1 week
  objectively measured with actigraph during one week
Sleep onset latency | 1 week
  objectively measured with actigraph during one week
Wake after sleep onset | 1 week
  objectively measured with actigraph during one week
Total sleep time | 1 week
  objectively measured with actigraph during one week
Self-reported sleep (Parental reported) | 1 week
  Subjectively measured sleep problems in smaller children, assessed by Child's Sleep Habits Questionnaire (CSHQ), assessed by the parents, referring to last week. consists of 33 items related to eight subscales; 1) Bedtime resistance, 2) Sleep onset delay, 3) Sleep duration, 4) Sleep anxiety, 5) Night wakings, 6) Parasomnias, 7) Sleep-disordered breathing, and 8) Daytime sleepiness. Each item is rated on a three-point scale: "usually" if the sleep behavior occurred five to seven times/week; "sometimes" for two to four times/week; and "rarely" for zero to one time/week. A higher score indicates more sleep problems
Self-reported sleep | 1 week
  Subjectively measured sleep problems in children, assessed by Insomnia Severity Index (ISI), children responding, referring to last week, comprises seven items for the children to respond to: 1) Severity of sleep-onset, 2) Sleep maintenance, 3) Early morning awakening, 4) Satisfaction with current sleep pattern, 5) Interference with daily functioning, 6) Noticeability of impairment attributed to the sleep problem, and 7) Level of distress caused by the sleep problem. Each item is rated on a five-point Likert scale ranging from "not at all" (scored at 0) to "extremely" (scored at 4). Total score ranges from 0 to 28, with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Parents' Health related quality of life | 1 day
  Assessed by EQ5D (among the parents), referring to this day. measuring the parents' health comprising five dimensions; 1) Mobility, 2) Self-care, 3) Usual activities, 4) Pain/discomfort, and 5) Anxiety/Depression. Each dimension is divided into three levels; No problems, Some or moderate problems, and extreme problems. In addition to the five dimensions, a 100-millimeter vertical Visual Analog Scale with endpoints of 100 means "best imaginable health state" and 0 means "worst imaginable health state is included. The total score ranges from 0 to 1 where a higher score indicates a better health-related quality of life.
Children's Health related quality of life | 1 day
  Assessed by EQ5D-y (among the children), referring to this day, comprises five items; 1) Walking about (mobility), 2) Looking after myself (self-care), 3) Doing usual activities (usual activities), 4) Having pain or discomfort (pain and discomfort), and 5) Feeling worried, sad or unhappy (anxiety and depression). Each item is divided into three levels; No problems, Some problems, and A lot of problems. The EQ-5D-Y also includes an easily understandable modified vertical Visual Analogue Scale of EQ-5D, where the respondent rates the overall health status with the endpoints from 0 (the worst health state the child can imagine and 100 (the best health state the child can imagine)
Children's general well-being | 1 day
  Assessed by Child Outcome Rating Scale (CORS), among the children, comprises four items where the child evaluates; 1) Me (How am I doing?), 2) Family (How are things in my family?), 3) School (How am I doing at school?), 4) Everything (How is everything going?). Each item is rated on a 100-millimeter Visual Analog Scale with smiling and sad faces as anchors.
Parent general well-being | 1 day
  Assessed by Outcome Rating Scale (ORS), among the parents assessment of the past week in four items; 1) Personal wellbeing, 2) Interpersonal relationships, 3) Social relations and, 4) Overall sense of well-being. Each item is rated on a 100-millimeter Visual Analog Scale with anchors from 0 (negative) to 100 (positive).
Anxiety | 1 day
  Assessed by short State-Trait Anxiety Inventory for children (short-STAI), includes six items.41 Each item is rated on a four-point Likert scale ranging with 1 = "not at all," 2 = "somewhat," 3, = "moderately", and 4 = "very much." The total score range from 6 to 24 points, with 6 points indicating no anxiety and 24 points indicating the highest level of anxiety.
ADHD symptoms | 1 week
  Assessed by The Swanson, Peland, and Nolan Scale (SNAP-IV), consists of 30 items and is divided into three subscales: inattention (nine items), hyperactivity/impulsivity (nine items), and oppositionality (eight items) and four supplementary questions regarding oppositionality (two questions) and ADHD (two questions). Items are rated on a four-point Likert scale range 0 = "not at all", 1 = "just a little", 2 = "quite a bit", and 3 = "very much". Items for inattention and hyperactivity/impulsivity can be combined to create a "combined ADHD" score.43 Higher scores represent more symptoms.
Family situation and parental mood | 1 week
  Assessed by Brief Child and Family Phone Interview (BCFPI), consists of 36 symptom items and another 36 items to assess function, adversity, and family stress grouped into 12 subscales. The subscale ´family situation' contains three items rated on a four-point Likert scale range 1 = never, 2 = sometimes, 3 = often, 4 =always. The subscale ´parental mood' contains six items based on the question "How often during the past week has the parent experienced…?" rated on a four-point scale; < 1 day, 1-2 days, 3-4 days, >5 days.
Cost effectiveness | 4 week
  Assessed by health economic aspects, such as absence from work, productivity, contact with health-care last four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Larsson, PhD, Principal Investigator — Halmstad University
Locations (1):
- Halmstad University, Halmstad, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsson I, Aili K, Nygren JM, Johansson P, Jarbin H, Svedberg P. SLEEP: intervention with weighted blankets for children with attention deficit hyperactivity disorder (ADHD) and sleep problems: study protocol for a randomised control trial. BMJ Open. 2022 Jan 4;12(1):e047509. doi: 10.1136/bmjopen-2020-047509. PMID 34983749